CLINICAL TRIAL: NCT02408757
Title: Multimodal Sonographic Monitoring of Cerebral Perfusion, Ventricle Seize and Optic Nerve Diameter During Weaning of Cerebrospinal Fluid Drainage Catheters: a Single Centre Observational Trial
Brief Title: Sonographic Monitoring of Weaning of Cerebrospinal Fluid Drainages
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: KEK 077/15
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Hydrocephalus
Keywords: ultrasound; cerebral perfusion; cerebrospinal fluid drainage
MeSH Terms: conditions — Hydrocephalus; Cerebrospinal Fluid Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: The study population consists of consecutive patients undergoing clamping of EVD/LD treated at the Departments of Neurosurgery or Intensive Care Medicine at the University Hospital Bern
  Interventions: Procedure: Sonographic monitoring

INTERVENTIONS:
Procedure: Sonographic monitoring — Sonographic monitoring during weaning of cerebrospinal fluid drainage catheters

SUMMARY:
As elaborated above only one study reported ultrasonographic changes of the width of the lateral ventricle during clamping of EVD/LD and indicated that ultrasound monitoring might be suitable. No firm data exists about the change of the width of the third ventricle, the diameter of the optic nerve or brain perfusion during clamping of the EVD/LD, although the width of these structures has been shown to depend on intracranial pressure. Ultrasonographic measurements of changes of the width of the third ventricle or the diameter of the optic nerve would have some advantages compared to the ultrasonographic assessments of the lateral ventricles. First, the width of the third ventricle can be measured easier and more reliable than the width of the lateral ventricles (better defined insonation plane and therefore higher repeatability of measurements) 3. Second, whereas assessments of the width of the side and third ventricles with ultrasound depend on the temporal bone windows (10 to 15% of patients have insufficient temporal bone windows), the measurement of the diameter of the optic nerve does not have this limitation and can therefore be performed in almost all patients. Hence, measurement of the diameter of the optic nerve would allow to overcome one major limitation of transcranial ultrasound. The latter limitation for transcranial ultrasound could also be minimized by the use of an ultrasound contrast agent (SonoVue®), but this was also not yet studied. The use of an ultrasound contrast agent would in addition allow to study changes of brain perfusion during clamping of EVD/LD.

DETAILED DESCRIPTION:
Background

Placement of a CSF drainage catheter (external ventricular drainage (EVD) or lumbar drainage (LD)) is a frequent neurosurgical emergency intervention. It is used in case of obstructive hydrocephalus as it can occur after e.g. intracerebral hemorrhage with intraventricular involvement, subarachnoid hemorrhage or traumatic brain injury but also in situations with reduced CSF resorption or increased CSF production (e.g. meningitis, ventriculitis). Furthermore, this technique can be used to monitor intracranial pressure. In all these situations, the EVD/LD can be used to reduce the elevated intracranial pressure during the acute phase. However, because of impairment of the Paccioni granulations by blood and its breakdown products, a continuing hydrocephalus may develop, leading to permanent necessity of CSF drainage. To evaluate the need for a permanent (implanted) drainage system (e.g. ventriculoperitoneal or ventriculoatrial shunt) attempts to clamp the EVD/LD are carried out during the subacute phase. Successful clamping is verified by absent increase of intracranial pressure, absent clinical deterioration and lack of ventricular enlargement on serial CT scans. The latter means that a first CT scan has to be performed before clamping of the drainage catheter (baseline examination) and again 24 hours after clamping of the drainage catheter. This leads to the need for repeated transportations of critically ill patients with possible harm of the patient, high costs, need for more staff and repeated exposure of the patient to radiation. Hence, a simple, repeatable, non-invasive, bedside tool for diagnosis of ventricular enlargement due to clamping of EVD/LD is strongly needed.

Transcranial ultrasound has become a widely used technique mainly for measuring arterial blood flow velocities. More recently, transcranial ultrasound has been also used to assess brain tissue, brain perfusion and ventricular size. The major advantages of ultrasound are its non-invasive character, the possibility for bedside application, low costs and safety (no X-ray exposure). Some studies have tried to use transcranial ultrasound for indirect assessment of intracranial pressure. As target structures for transcranial ultrasound either the lateral ventricles, the third ventricle or the diameter of the optic nerve were used. All studies could demonstrate a correlation between the width of the lateral or third ventricle or the diameter of the optic nerve with intracranial pressure. To the investigators' knowledge, only one study assessed the change of the width of the lateral ventricles during clamping of EVD/LD.

To summarize, a bedside method for assessment of changes of ventricle width/diameter of the optic nerve during clamping of EVD/LD is urgently needed and would facilitate the procedure, higher patient safety and lower costs. By now, there are some promising ultrasound methods (transcranial ultrasound with or without contrast enhancing agent to determine the width of the side and third ventricle, diameter of the optic nerve), which might substitute repeated CT scans but have not been evaluated for monitoring clamping of EVD/LD.

Objective

The investigators hypothesize that clamping of EVD/LD can be monitored using repeated bedside ultrasound examinations instead of repeated CT scans. The purpose of this study is to investigate if a multimodal approach consisting of ultrasonographic determination of changes of the width of the third and the side ventricles as well as the diameter of the optic nerve can be used to screen for ventricle enlargement during clamping of EVD/LD. To this end, the investigators will compare a classifier based on ultrasound with the clinical decision based on CT.

Methods

The study consists of two additional ultrasonographic examinations . The standard treatment of patients undergoing clamping of EVD/LD is not affected by the study. The first ultrasonographic examination is performed in parallel to the baseline CT scan (either immediately before or after the CT scan) before clamping of the EVD/LD. The second ultrasound is made 24 hours after clamping of the EVD/LD in parallel to the follow-up CT Scan (either immediately before or after the CT scan). The examinations will be made bedside in the supine position on the ward where the patient is treated.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of patient or relative and statement of independent physician
* Patient treated with EVD or LD undergoing clamping of EVD/LD
* Age ≥18 ≤ 80 years

Exclusion Criteria

* Pregnancy and breastfeeding
* Acute coronary syndromes, severe ischemic heart disease (requiring revascularisation), severe aortic and mitral valve disease, severe congestive heart failure (NYHA >III/IV)
* Severe pulmonary or renal dysfunction
* Known allergy or adverse reaction to contrast material

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of consecutive patients undergoing clamping of EVD/LD treated at the Departments of Neurosurgery or Intensive Care Medicine at the University Hospital Bern
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
binary classification of patients in terms of change of width of cerebrospinal fluid spaces by ultrasound | 24 hours after clamping of EVD/LD

SECONDARY OUTCOMES:
change of width of the third ventricle measured with transcranial ultrasound without ultrasound contrast agent | 24 hours after clamping of EVD/LD
change of width of the third ventricle measured with transcranial ultrasound with ultrasound contrast agent | 24 hours after clamping of EVD/LD
change of width of the lateral ventricles measured with transcranial ultrasound without ultrasound contrast agent | 24 hours after clamping of EVD/LD
change of diameter of the optic nerve | 24 hours after clamping of EVD/LD
change of width of the third ventricle in the CT scan | 24 hours after clamping of EVD/LD
change of width of the lateral ventricles in the CT scan | 24 hours after clamping of EVD/LD
change of brain perfusion in the brain regions adjacent to the third ventricle | 24 hours after clamping of EVD/LD

CONTACTS AND LOCATIONS:
Overall Officials: Werner Z'Graggen, MD, Principal Investigator — Department of Neurosurgery, University Hospital Bern
Locations (1):
- Inselspital Bern, Bern, Switzerland

REFERENCES:
- [Background] Voigt LP, Pastores SM, Raoof ND, Thaler HT, Halpern NA. Review of a large clinical series: intrahospital transport of critically ill patients: outcomes, timing, and patterns. J Intensive Care Med. 2009 Mar-Apr;24(2):108-15. doi: 10.1177/0885066608329946. Epub 2009 Feb 2. PMID 19188270
- [Background] Waydhas C. Intrahospital transport of critically ill patients. Crit Care. 1999;3(5):R83-9. doi: 10.1186/cc362. Epub 1999 Sep 24. PMID 11094486
- [Background] Becker G, Bogdahn U, Strassburg HM, Lindner A, Hassel W, Meixensberger J, Hofmann E. Identification of ventricular enlargement and estimation of intracranial pressure by transcranial color-coded real-time sonography. J Neuroimaging. 1994 Jan;4(1):17-22. doi: 10.1111/jon19944117. PMID 7907896
- [Background] Bolesch S, von Wegner F, Senft C, Lorenz MW. Transcranial ultrasound to detect elevated intracranial pressure: comparison of septum pellucidum undulations and optic nerve sheath diameter. Ultrasound Med Biol. 2015 May;41(5):1233-40. doi: 10.1016/j.ultrasmedbio.2014.12.023. Epub 2015 Jan 28. PMID 25638313
- [Background] Kiphuth IC, Huttner HB, Struffert T, Schwab S, Kohrmann M. Sonographic monitoring of ventricle enlargement in posthemorrhagic hydrocephalus. Neurology. 2011 Mar 8;76(10):858-62. doi: 10.1212/WNL.0b013e31820f2e0f. Epub 2011 Feb 2. PMID 21288979
- [Background] Jungehulsing GJ, Brunecker P, Nolte CH, Fiebach JB, Kunze C, Doepp F, Villringer A, Schreiber SJ. Diagnostic transcranial ultrasound perfusion-imaging at 2.5 MHz does not affect the blood-brain barrier. Ultrasound Med Biol. 2008 Jan;34(1):147-50. doi: 10.1016/j.ultrasmedbio.2007.07.006. Epub 2007 Sep 14. PMID 17854981
- [Background] Engelhardt M, Hansen C, Eyding J, Wilkening W, Brenke C, Krogias C, Scholz M, Harders A, Ermert H, Schmieder K. Feasibility of contrast-enhanced sonography during resection of cerebral tumours: initial results of a prospective study. Ultrasound Med Biol. 2007 Apr;33(4):571-5. doi: 10.1016/j.ultrasmedbio.2006.10.007. PMID 17337111
- [Background] Kopp R, Zurn W, Weidenhagen R, Meimarakis G, Clevert DA. First experience using intraoperative contrast-enhanced ultrasound during endovascular aneurysm repair for infrarenal aortic aneurysms. J Vasc Surg. 2010 May;51(5):1103-10. doi: 10.1016/j.jvs.2009.12.050. PMID 20420978
- [Background] Shah AJ, Callaway M, Thomas MG, Finch-Jones MD. Contrast-enhanced intraoperative ultrasound improves detection of liver metastases during surgery for primary colorectal cancer. HPB (Oxford). 2010 Apr;12(3):181-7. doi: 10.1111/j.1477-2574.2009.00141.x. PMID 20590885
- [Background] Wu H, Lu Q, Luo Y, He XL, Zeng Y. Application of contrast-enhanced intraoperative ultrasonography in the decision-making about hepatocellular carcinoma operation. World J Gastroenterol. 2010 Jan 28;16(4):508-12. doi: 10.3748/wjg.v16.i4.508. PMID 20101780
- [Background] Bokor D, Chambers JB, Rees PJ, Mant TG, Luzzani F, Spinazzi A. Clinical safety of SonoVue, a new contrast agent for ultrasound imaging, in healthy volunteers and in patients with chronic obstructive pulmonary disease. Invest Radiol. 2001 Feb;36(2):104-9. doi: 10.1097/00004424-200102000-00006. PMID 11224758
- [Background] Piscaglia F, Bolondi L; Italian Society for Ultrasound in Medicine and Biology (SIUMB) Study Group on Ultrasound Contrast Agents. The safety of Sonovue in abdominal applications: retrospective analysis of 23188 investigations. Ultrasound Med Biol. 2006 Sep;32(9):1369-75. doi: 10.1016/j.ultrasmedbio.2006.05.031. PMID 16965977